CLINICAL TRIAL: NCT02442752
Title: A Phase 1, Randomized, Open-Label, Parallel-Design, Multicenter Study to Evaluate the Pharmacokinetics, Safety, and Pharmacodynamics of Dexlansoprazole Delayed-Release Capsules in Infants Aged 1 to 11 Months With Acid-Related Diseases
Brief Title: Phase 1 Dexlansoprazole Delayed-Release Capsules for Acid-Related Disorders in Infants Aged 1 to 11 Months
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn: Business decision (no enrollment)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-390MR_108; 2014-001642-16 (EudraCT Number); U1111-1162-4853 (Registry Identifier: WHO); 153300410A0065 (Registry Identifier: NREC)
Record Dates: First submitted 2015-05-09; First posted 2015-05-13 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Pediatric Gastroesophageal Reflux Disease
Keywords: Drug therapy
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen A: Dexlansoprazole 10 mg (Experimental): Dexlansoprazole 10 mg, delayed-release capsules, orally, once daily for 8 weeks.
  Interventions: Drug: Dexlansoprazole
- Regimen B: Dexlansoprazole 15 mg (Experimental): Dexlansoprazole 15 mg, delayed-release capsules, orally, once daily for 8 weeks.
  Interventions: Drug: Dexlansoprazole
- Regimen C: Dexlansoprazole 20 mg (Experimental): Dexlansoprazole 20 mg, delayed-release capsules, orally, once daily for 8 weeks.
  Interventions: Drug: Dexlansoprazole
- Regimen D: Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg, delayed-release capsules, orally, once daily for 8 weeks.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole capsules
  Other Names: TAK-390MR

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) and pharmacodynamics (PD) [after daily administration for 7 days] and safety [after daily administration for 8 weeks] of dexlansoprazole in pediatric participants aged 1 to 11 months, inclusive, with acid-related diseases.

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. Dexlansoprazole is being tested to find a safe and well-tolerated dose and to assess how dexlansoprazole is processed by the body in infants aged 1 to 11 months. This study will look at side effects and lab results in infants who take dexlansoprazole.

The study will enroll approximately 24 participants. Participants will be randomly assigned to 1 of the 4 treatment groups based on body weight and age:

* Dexlansoprazole 10 mg
* Dexlansoprazole 15 mg
* Dexlansoprazole 20 mg
* Dexlansoprazole 30 mg

Participants who weigh <3.4 kg will not be enrolled. Participants ≤ 10 weeks of age with a body weight of ≥ 3.4 kg will initially receive Regimen A (dexlansoprazole delayed-release 10 mg capsules). Randomization for participants > 10 weeks of age will be stratified by weight group. Participants whose baseline weight is ≥ 3.4 kg but < 4.1 kg will be assigned to receive Regimen A or Regimen B (dexlansoprazole delayed-release 10 or 15 mg capsules as an initial dose) in a ratio of 1:1. Participants whose weight is ≥ 4.1 kg but < 6.2 kg will be assigned to receive Regimens B or C (dexlansoprazole delayed-release 15 or 20 mg capsules as an initial dose) in a ratio of 1:1. Participants whose weight is ≥ 6.2 kg will be assigned to receive Regimen B, C, or D (dexlansoprazole delayed-release 15, 20, or 30 mg capsules as an initial dose) in a ratio of 1:1:2.

All participants will be administered 1 capsule of dexlansoprazole in the morning at the same time each day throughout the study. The study medication may be administered to the participants by opening a capsule and sprinkling the granules on 1 tablespoon of applesauce or pureed apples, or mixing the capsule granules with about 20 mL of water. The food-granule mixture should be administered immediately. The water mixed with the granules will be administered via an oral syringe into the mouth immediately. The granules should not be chewed in mouth. The food or liquid used for administering the study medication should be recorded for Days 1 through Confinement Day 1. The parents of all participants will be asked to record dosing information, the food or liquid used for administering the study medication (Day 1 through Confinement Day 1), food intake, and episodes of vomiting in a diary from Day 2 until the day before Confinement Day 1 (Day 5 to 9).

This multicenter trial will be conducted worldwide. The overall time to participate in this study is up to 114 days. Participants will make multiple visits to the clinic, including two 2-day visits that may require confinement to the clinic, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to any study-specific procedures being performed and after having the study fully explained and all questions answered, the informed consent form (ICF) must be signed and dated by parent(s) or legal guardian(s). The Screening Period starts at the time of consent.
2. Is a male or female infant 1 to 11 months old, inclusive, on Day 1. Infants who were born prematurely must be ≥ 45 weeks old based on corrected gestational age.
3. At the Initial Screening and Day -1 visits, participant must have body weight percentile-for-age within the 5th through 95th percentile by age, inclusive, as determined by the World Health Organization (WHO) growth chart.
4. Must be ≥ 3.4 kg at the Screening and Day -1 visits.
5. Participants who take a prescription or nonprescription proton pump inhibitor (PPI), histamine-2 receptor antagonists(H2RA), sucralfate, or antacids on a regular or as required basis must agree to discontinue use at Day -1 (except cimetidine, which must be discontinued 28 days prior to Day -1) or other acid suppression therapy, and agree to discontinue use throughout the study.
6. Must have endoscopically proven erosive esophagitis (EE), a history of EE, and/or 1 or more of the following underlying conditions that predispose the participant to chronic gastroesophageal reflux disease (GERD) and EE: moderate to severe neurologic impairment, repaired esophageal atresia, hiatal hernia, cystic fibrosis, bronchopulmonary dysplasia, or end-stage renal disease.
7. Except for participants with EE, a history of EE, or repaired esophageal atresia, participants have:

   * Received prior PPI therapy or other acid suppression therapy for a minimum of 2 weeks during any time in the past with symptomatic response and have demonstrated a recurrence of symptoms following at least 1 attempted withdrawal of PPI therapy or other acid suppression therapy AND
   * Have undergone esophageal pH monitoring in the recent past to document that their symptoms are due to acid-mediated disease.
8. Must be able to ingest study medication granules sprinkled on 1 tablespoon of applesauce or pureed apples, or as a mixture of granules in water administered via an oral syringe.
9. Must be at least 7 days post-surgery by dosing on Day 1 and have no anticipated need for surgery during the study.
10. Screening laboratory samples must be collected Day -7 to Day -2) and the results must be within the range expected for this infant population (except gastrin results as those results will be available after Day 1). The laboratory results should indicate no clinically significant (CS) abnormality in chemistry (including electrolytes, blood urea nitrogen [BUN]), creatinine, glucose, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin), hematology (complete blood cell count, including differential), and urinalysis parameters (if standard of care).

Exclusion Criteria:

1. Has evidence of cardiovascular, pulmonary, central nervous system, hepatic, hematopoietic, renal, metabolic, endocrine or gastrointestinal disease, or serious allergy, asthma, or allergic skin rash that suggests clinically significant, uncontrolled underlying disease or condition (other than the disease being studied and/or identified as the main criterion for inclusion), that may impact the ability of the participant to participate or potentially may confound the study results.
2. Has known history of or current presence of peptic ulcers or gastrointestinal bleeding (hematemesis, hematochezia).
3. Has poor venous access or any contraindication to blood sampling.
4. Has known history of eosinophilic gastroenteropathy, or a coexisting disease affecting the esophagus, including esophageal varices, viral or fungal infection, or esophageal stricture, history of radiation therapy or cryotherapy to the esophagus, and caustic or physiochemical trauma such as sclerotherapy to the esophagus.
5. Has active malabsorption syndrome, cow's milk intolerance, milk protein allergy, or celiac disease.
6. Has any finding in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of a disease that might interfere with the conduct of the study or that would contraindicate taking dexlansoprazole delayed-release capsules or a similar drug in the same class (ie, a PPI).
7. Has a known hypersensitivity to any PPI or any component of the formulation of dexlansoprazole delayed-release capsules.
8. Is required to take excluded medications or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study evaluation period.
9. Has a history of malignant disease.
10. Has a known history of infection with the human immunodeficiency virus.
11. Has lost > 10% of the total blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study medication.
12. Has consumed Excluded Medications and Dietary Products during the time periods listed, or parent(s) or legal guardian(s) is unwilling to agree to participant abstaining from products while participating in the study.
13. Has participated in a study of an investigational agent (including dosing or follow-up) within 30 days prior to Screening.
14. Has a Screening Visit laboratory value that the principal investigator and sponsor consider to be clinically significant.
15. Has creatinine > 1.5 mg/dL, ALT and/or AST > 2 times the upper limit of normal (ULN), or total bilirubin > 2.0 mg/dL with AST/ALT elevated above the limits of normal values.
16. The participant or parent/legal guardian is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study or may consent under duress.
17. Parent/legal guardian, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.
18. Has any congenital anomaly of the upper gastric intestinal tract that might interfere with gastrointestinal motility, pH, or absorption, or has an active or known history of necrotizing enterocolitis that has been surgically corrected.
19. Has clinical evidence of acute sepsis. Infants on chronic antibiotics who are otherwise clinically stable may be enrolled in the study at the discretion of the investigator.
20. Has received a vaccine within 48 hours prior to dosing on Day 1.
21. Has used intravenous or oral antifungal agents within the 7 days prior to Day -1.
22. Has used mucosal protective agent (eg, sucralfate) within 6 hours prior to dosing on Day 1.

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Dexlansoprazole | Confinement Day 1 (Between Day 5 and Day 9) Pre-dose, and at multiple timepoints (up to 12 hours) post-dose
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Area Under the Plasma Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUCt) of Dexlansoprazole | Confinement Day 1 (Between Day 5 and Day 9) Pre-dose, and at multiple timepoints (up to 12 hours) post-dose
  Area under the plasma concentration versus time curve from time zero to the time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time 0 to Time tau [AUCtau)] for Dexlansoprazole | Confinement Day 1 (Between Day 5 and Day 9) Pre-dose, and at multiple timepoints (up to 12 hours) post-dose
  Area under the plasma concentration-time curve from time 0 to time tau, where tau is the length of the dosing interval.
Dose Normalized Maximum Observed Plasma Concentration (Cmax/dose) of Dexlansoprazole | Confinement Day 1 (Between Day 5 and Day 9) Pre-dose, and at multiple timepoints (up to 12 hours) post-dose
  Dose normalized maximum observed plasma concentration (Cmax/dose) is the peak plasma concentration of a drug after administration obtained directly from the plasma concentration-time curve, divided by the administered dose in milligrams.
Dose Normalized Area Under the Plasma Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUCt/dose) of Dexlansoprazole | Confinement Day 1 (Between Day 5 and Day 9) Pre-dose, and at multiple timepoints (up to 12 hours) post-dose
  Area under the plasma concentration versus time curve from time zero to the time of the last quantifiable concentration divided by the administered dose in milligrams.
Dose Normalized Area Under the Plasma Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUCt/dose) of Dexlansoprazole | Confinement Day 1 (Between Day 5 and Day 9) Pre-dose, and at multiple timepoints (up to 12 hours) post-dose
  Area under the plasma concentration-time curve during a dosing interval, where tau is the length of the dosing interval, divided by the administered dose in milligrams.
Change from Baseline in Percent of Time with Intragastric pH>4 | Baseline and Confinement Day 1(Between Day 5 and Day 9) [up to 24 hours post-dose]
  Intragastric pH will be measured approximately every 2 to 4 seconds, based on the pH recorder used for the measurement, for a 24-hour period. Fifteen minute medians are calculated and the percent of time pH is greater than 4 is calculated for the 24 hour period.
Change from Baseline in Mean 24-Hour Intragastric pH | Baseline and Confinement Day 1(Between Day 5 and Day 9) [up to 24 hours post-dose]
  Intragastric pH will be measured approximately every 2 to 4 seconds, based on the pH recorder used for the measurement, for a 24-hour period. Fifteen minute medians are calculated and the mean pH is calculated for the 24 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (22):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Michigan Pediatric GI Center, Flint, Michigan
  - Promedica Toledo Children's Hospital, Toledo, Ohio
  - Cook Children's Medical Center, Fort Worth, Texas
- Israel (4):
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Assaf Harofeh M.C, Rishon LeZiyyon
- Italy (4):
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Umberto I Pol. di Roma-Universita di Roma La Sapienza, Roma
  - Ospedale Pediatrico Bambino Gesu, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
- Mexico (3):
  - Centro de Investigacion Clinica Acelerada, S.C., Mexico City, Mexico City
  - Centro de Investigacion Clinica Chapultepec S.A. de C.V., Morelia, Michoacán
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
- Poland (5):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Uniwersytecki Szpital Dzieciecy w Lublinie, Lublin
  - Szpital Wojewodzki nr 2 w Rzeszowie, Rzeszów
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw